CLINICAL TRIAL: NCT03227042
Title: A Prospective Natural History Study of Mucopolysaccharidosis Type IIIB (MPS IIIB)
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Allievex Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: 250-902
Record Dates: First submitted 2017-07-11; First posted 2017-07-24 (Actual); Last update posted 2022-10-26 (Actual); Status verified 2022-10

CONDITIONS: Mucopolysaccharidosis Type IIIB
Keywords: Sanfilippo Syndrome Type B; MPS IIIB; MPS 3 B
MeSH Terms: conditions — Mucopolysaccharidosis III

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a natural history study for children up to 18 years of age who have been diagnosed with Mucopolysaccharidosis Type IIIB (MPS IIIB, also known as Sanfilippo Syndrome Type B). Mucopolysaccharidosis type IIIB is a severe neurodegenerative disorder. The information gathered from this trial may help inform the design and interpretation of subsequent interventional studies. No clinical intervention or study drug is provided by Allievex in this study.

ELIGIBILITY:
Inclusion Criteria:

* Have deficient NAGLU enzyme activity at Baseline. Blood for NAGLU enzyme activity will be collected and analyzed centrally.
* Is up to 18 years of age
* Written informed consent from parent or legal guardian and assent from subject, if required
* Has the ability to comply with protocol requirements, in the opinion of the investigator

Exclusion Criteria:

* Has another neurological illness that may have caused cognitive decline (e.g., trauma, meningitis, or hemorrhage) before study entry
* Has received stem cell, gene therapy, or enzyme replacement therapy for MPS IIIB
* Has received any investigational medication within 30 days prior to the Baseline visit or is scheduled to receive any investigational drug during the course of the study
* Has a medical condition or extenuating circumstance that, in the opinion of the investigator, might compromise the subject's ability to comply with protocol requirements, the subject's wellbeing or safety, or the interpretability of the subject's clinical data.
* Is currently participating in another natural history study

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Males and Females with a documented diagnosis of MPSIIIB
Sampling Method: Non-Probability Sample
Enrollment: 44 (Actual)
Dates: Start 2017-11-16 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Neurocognitive function | Baseline + every 24 weeks for up to 240 weeks
  A neurodevelopmental assessment will be performed using standardized developmental tests to provide quantifiable measures of neurocognitive function.
Behavioral function | Baseline + every 24 weeks for up to 240 weeks
  Disease-related behaviors will be assessed using an MPS IIIB specific behavior rating scale.
Quality of Life Tests | Baseline + every 24 weeks for up to 240 weeks
  Multiple QoL tools will be used to capture physical, mental, and social well-being of the patient as well as to examine the impact of the patient's disease on the parent/guardian and family.
Sleep habits | Baseline + every 24 weeks for up to 240 weeks
  Patient sleep habits will be assessed using Children's Sleep Habits Questionnaires (CSHQ).
Disease-specific Biomarkers | Baseline + every 24 weeks for up to 240 weeks
  Urine sample for glycosaminoglycans (GAGs) and creatinine.
Biochemical, Molecular, Cellular and Genetic Markers of Disease Burden | Once (at baseline visit)
  Blood and urine samples will be used to evaluate biochemical, molecular cellular, and genetic/genomic aspects of MPS IIIB.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, MD, Study Director — Allievex Medical Monitor
Locations (9):
- UCSF Benioff Children's Hospital Oakland, Oakland, California, United States
- Hospital Universitario Austral, Pilar, Argentina
- Murdoch Childrens Research Institute and Royal Children's Hospital, Melbourne, Victoria, Australia
- Medical Genetics Service/HCPA, Department of Genetics/UFRGS, Pôrto Alegre, Rio Grande do Sul, Brazil
- Fundación Cardio Infantil - Instituto de Cardiología, Bogotá, Colombia
- University Medical Center Hamburg-Eppendorf, Hamburg, Germany
- Hospital Clínico Universitario de Santiago, Santiago de Compostela, A Coruña, Spain
- MacKay Memorial Children's Hospital, Taipei, Taiwan
- Gazi University Faculty of Medicine, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Okur I, Ezgu F, Giugliani R, Muschol N, Koehn A, Amartino H, Harmatz P, de Castro Lopez MJ, Couce ML, Lin SP, Batzios S, Cleary M, Solano M, Peters H, Lee J, Nestrasil I, Shaywitz AJ, Maricich SM, Kuca B, Kovalchin J, Zanelli E. Longitudinal Natural History of Pediatric Subjects Affected with Mucopolysaccharidosis IIIB. J Pediatr. 2022 Oct;249:50-58.e2. doi: 10.1016/j.jpeds.2022.06.005. Epub 2022 Jun 13. PMID 35709957